CLINICAL TRIAL: NCT04976946
Title: Protocol for CAMUS Delphi Study: A Consensus on Reporting of Complications After Urological Surgeries
Brief Title: Protocol for CAMUS Delphi Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Other Study IDs: 2020.046
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Complications; Urogenital, Postprocedural

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Urologists: Local and international consultant Urologists and accredited Urology trainees.
  Interventions: Other: Comprehensive questionnaire
- Anaesthetists: Local and international consultant anaesthetists. Critical care physicians who are primarily Urological anaesthetists or have experience in complication reporting will be targeted.
  Interventions: Other: Comprehensive questionnaire
- ICU specialists: Local and international consultant ICU specialists. Critical care physicians who are primarily Urological focused or have experience in complication reporting will be targeted.
  Interventions: Other: Comprehensive questionnaire

INTERVENTIONS:
Other: Comprehensive questionnaire — Multi-staged, international Delphi study that aims to establish criteria for standardised complication reporting in Urology.

SUMMARY:
Multi-staged, international Delphi study that aims to establish criteria for standardised complication reporting in Urology.

DETAILED DESCRIPTION:
The CAMUS Delphi Study: A Consensus on Reporting of Complications After Urological Surgeries is a multi-staged, international Delphi study that aims to establish criteria for standardised complication reporting in Urology. The initial survey consists of a 12-part questionnaire that will aim to reach consensus on a wide range of contentious issues in Urological surgery using the frameworks of both the established Clavien-Dindo Classification (CDC) and the new CAMUS Classification.

To ensure comprehensive and comparable complication reporting across centres worldwide, a conclusive uniform language for reporting complications must be created and subsequently integrated. Accurate reporting will allow for more precise allocation of resources, improve unit efficiency, and reduce healthcare burden, while providing clinicians with a better understanding of intra- and post-operative morbidity. If a comprehensive, homogenous reporting construct is integrated worldwide, the potential to build and develop a universal database with complications from all centres around the world will surely provide invaluable data to create new guidelines and recommendations, ultimately improving patient counselling and surgical quality of care.

ELIGIBILITY:
Inclusion Criteria:

* Local and international consultant Urologists, accredited Urology trainees, consultant Anaesthetists and consultant ICU specialists will be invited to complete the survey. Critical care physicians who are primarily Urological anaesthetists or have experience in complication reporting will be targeted.

Exclusion Criteria:

* All other specialists that do not meet the inclusion criteria.
* Under 18 years of age.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Local and international consultant Urologists, accredited Urology trainees, consultant Anaesthetists and consultant ICU specialists will be invited to complete the survey. Critical care physicians who are primarily Urological anaesthetists or have experience in complication reporting will be targeted. Must be over the age of 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Standardised complication reporting in Urology | 6 months
  Establish criteria for standardised complication reporting in Urology

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Furrer, MD, Principal Investigator — Melbourne Health
Locations (1):
- The Royal Melbourne Hospital, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: Undecided